CLINICAL TRIAL: NCT02439632
Title: A Multi-center, Randomized, Double-blind, Double-dummy Clinical Study to Evaluate the Safety and Efficacy of Prulifloxacin Film-coated Tablet for the Treatment of Acute Uncomplicated Lower Urinary Tract Infection With Levofloxacin Hydrochloride Tablet as Active Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prulifloxacin aulut ZK-004
Record Dates: First submitted 2014-06-04; First posted 2015-05-12 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-05

CONDITIONS: Acute Lower Urinary Tract Infection
MeSH Terms: interventions — prulifloxacin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- prulifloxacin (Experimental): Prulifloxacin film-coated tablet : 600 mg/tablet, oral administration of a single tablet.
  Placebo of levofloxacin hydrochloride tablet without active components.
  Interventions: Drug: prulifloxacin; Drug: Levofloxacin Placebo
- Levofloxacin (Active Comparator): Levofloxacin hydrochloride tablet 250 mg/tablet, oral administration of a tablet daily for a total of 3 days.
  Placebo of prulifloxacin film-coated tablet, without active components.
  Interventions: Drug: Levofloxacin; Drug: Prulifloxacin Placebo

INTERVENTIONS:
Drug: prulifloxacin
  Arms: prulifloxacin
Drug: Levofloxacin — Levofloxacin hydrochloride tablet 250 mg/tablet, oral administration of a tablet daily for a total of 3 days.
  Arms: Levofloxacin
Drug: Prulifloxacin Placebo — Placebo of prulifloxacin film-coated tablet without active components.
  Arms: Levofloxacin
Drug: Levofloxacin Placebo — Placebo of levofloxacin hydrochloride tablet without active components.
  Arms: prulifloxacin

SUMMARY:
prulifloxacin is not inferior to levofloxacin hydrochloride in treating acute uncomplicated lower urinary tract infection in chinese

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 ~ 65 years old;
2. Presence at least two of the following clinical signs and symptoms of acute uncomplicated lower urinary tract infection: dysuria, frequency, urgency and suprapubic pain) with onset of symptoms ≤ 72 hours prior to study entry;
3. With pyuria: WBC > 10/mm3 in unspun urine examined in a counting chamber or WBC > 5/hp [or the Upper laboratory Norm (UNL)] in the resuspended sediment of a centrifuged aliquot of urine (or the UNL);
4. Patient is willing to participate in the study and gives the signature of informed consent form;

Exclusion Criteria:

1. Presence of clinical signs and symptoms suggestive of pyelonephritis or complicated urinary tract infection (e.g., fever > 37.5°C, chills, flank pain), or with factors associated with complicated urinary tract infections such as presence of an indwelling catheter or urologic abnormalities;
2. Women who are pregnant, nursing or plan to become pregnant in the near future (i.e., in three months). Women of childbearing potential (post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential) must have a negative serum pregnancy test at screening and must be willing to use an acceptable method of contraception to avoid pregnancy throughout the study. Acceptable methods of contraception include tubal ligation, oral contraceptive, barrier methods (intra-uterine device, diaphragm, female condom, male condom);
3. Three or more episodes of acute uncomplicated UTI in the past 12 months;
4. Patients with overactive bladder;
5. Patients are hypersensitive to quinolones or with allergic constitution;
6. Administration of xanthines, fenbufen, antibiotics or antibacterials within the two previous weeks;
7. Patients with severe condition which need combination with other antibacterial agents or corticosteroids during the study;
8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, Inflammatory bowel disease, lactose intolerance, or malabsorption syndrome)
9. Patients with severe liver or kidney disease, defined as serum ALT and AST ≥ 2.5 x ULN and creatinine ≥ 1.5 x ULN;
10. Patients with severe heart disease or Q-T prolongation indicated by 12-lead ECG, or arrhythmia or acute myocardial ischemia;
11. WBC < 3.6 × 109/L or neutrophil < 1.8 × 109/L, and/or platelets < 90 × 109/L at screening;
12. Patients with central nervous system disease or convulsion history, and/or with mental status unable to coordinate;
13. Patients with malignant tumor or other severe background disease;
14. Patients with severe immunodeficiency;
15. Patients with a history of tendinopathy or who are currently having the disease, including tendinitis and tendon rupture;
16. Patients treated with experimental drugs in the previous 4 weeks or currently;
17. Considered inappropriate for the study by investigators, including patients who are unable or unwilling to show compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The efficacy of prulifloxacin film-coated tablet was meaured by the number of patient have been cured | 3 days
  600mg single dose prolifloxacin is not inferior to Levoflxacin on low urine infection in Chinese

SECONDARY OUTCOMES:
The safety of prulifloxacin film-coated tablet was measured by the number fo AE and SAE | 3 days and 28 days
  1. The susceptibility of infecting strains to prulifloxacin;
  2. The rate of return to normal of WBC (white blood cell) in urine in treatment and control group
  3. The safety and tolerability of prulifloxacin in adult patients with acute lower urinary tract infection

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Medical Union Hospital, Beijing, China